CLINICAL TRIAL: NCT00716976
Title: A Randomized Phase III Study of Sodium Thiosulfate for the Prevention of Cisplatin-Induced Ototoxicity in Children
Brief Title: Sodium Thiosulfate in Preventing Hearing Loss in Young Patients Receiving Cisplatin for Newly Diagnosed Germ Cell Tumor, Hepatoblastoma, Medulloblastoma, Neuroblastoma, Osteosarcoma, or Other Malignancy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ACCL0431; COG-ACCL0431 (Other: Children's Oncology Group); CDR0000588655 (Other: Clinical Trials.gov)
Record Dates: First submitted 2008-07-15; First posted 2008-07-16 (Estimated); Results first posted 2017-06-01 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2021-07

CONDITIONS: Brain Tumor; Central Nervous System Tumor; Childhood Germ Cell Tumor; Extragonadal Germ Cell Tumor; Liver Cancer; Neuroblastoma; Ototoxicity; Ovarian Cancer; Sarcoma
Keywords: ototoxicity; childhood central nervous system germ cell tumor; childhood extracranial germ cell tumor; childhood extragonadal germ cell tumor; childhood malignant testicular germ cell tumor; childhood malignant ovarian germ cell tumor; childhood teratoma; childhood medulloblastoma; disseminated neuroblastoma; regional neuroblastoma; localized resectable neuroblastoma; localized unresectable neuroblastoma; stage 4S neuroblastoma; localized osteosarcoma; metastatic osteosarcoma; childhood hepatoblastoma; stage I childhood liver cancer; stage II childhood liver cancer; stage III childhood liver cancer; stage IV childhood liver cancer
MeSH Terms: conditions — Brain Neoplasms; Central Nervous System Neoplasms; Liver Neoplasms; Neuroblastoma; Ototoxicity; Ovarian Neoplasms; Sarcoma; Testicular Neoplasms; Ovarian Germ Cell Cancer; Teratoma; Medulloblastoma; Osteosarcoma; Hepatoblastoma | interventions — sodium thiosulfate; Restraint, Physical

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- STS Arm (sodium thiosulfate treatment) (Experimental): Patients receive sodium thiosulfate IV (dosage 16 g/m2 or 533 mg per kg for patients whose therapeutic protocol administers cisplatin on a per kg basis due to young age or small body) over 15 minutes beginning 6 hours after the completion of each cisplatin infusion. Treatment with sodium thiosulfate continues until the completion of cisplatin therapy.
  Interventions: Drug: sodium thiosulfate; Procedure: examination
- Observation Arm (No sodium thiosulfate treatment) (Experimental): Patients do not receive sodium thiosulfate.
  Interventions: Procedure: examination

INTERVENTIONS:
Drug: sodium thiosulfate — Given IV
  Other Names: ADH300001; Disodium Thiosulfate Pentahydrate; Na Thiosulfate; Sodium Hyposulfite; Sodium Thiosulphate; Thiosulfuric Acid; Disodium Salt; Pentahydrate; Versiclear; NSC# 45624; IND#72877
  Arms: STS Arm (sodium thiosulfate treatment)
Procedure: examination — Patients undergo audiological assessments periodically

SUMMARY:
RATIONALE: Sodium thiosulfate may reduce or prevent hearing loss in young patients receiving cisplatin for cancer. It is not yet known whether sodium thiosulfate is more effective than no additional treatment in preventing hearing loss.

PURPOSE: This randomized phase III trial is studying sodium thiosulfate to see how well it works in preventing hearing loss in young patients receiving cisplatin for newly diagnosed germ cell tumor, hepatoblastoma, medulloblastoma, neuroblastoma, osteosarcoma, or other malignancy.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To compare the efficacy of sodium thiosulfate vs observation in preventing hearing loss in young patients receiving cisplatin for the treatment of newly diagnosed germ cell tumor, hepatoblastoma, medulloblastoma, neuroblastoma, osteosarcoma, or other malignancy.

Secondary

* To compare the mean change in hearing thresholds for key frequencies in these patients.
* To compare the incidences of cisplatin-related grade 3 and 4 nephrotoxicity and grade 3 and 4 cytopenia in these patients.
* To compare the event-free survival and overall survival of these patients.
* To evaluate the association of two key gene mutations (TPMT and COMT) with the development of cisplatin-induced hearing loss in these patients.

OUTLINE: This is a multicenter study. Patients are stratified according to prior cranial radiation (yes vs no), age (< 5 years vs ≥ 5 years) and duration of cisplatin infusion (< 2 hours vs ≥ 2 hours). Patients are randomized to 1 of 2 arms.

* Arm I (sodium thiosulfate): Patients receive sodium thiosulfate IV over 15 minutes beginning 6 hours after the completion of each cisplatin infusion. Treatment with sodium thiosulfate continues until the completion of cisplatin therapy.
* Arm II (observation): Patients do not receive sodium thiosulfate.

Patients undergo audiological assessment at baseline, prior to each course of cisplatin, and then at 4 weeks and 1 year after the last course of cisplatin or other cancer treatment. Some patients may undergo saliva collection for DNA studies.

After completion of study, patients are followed periodically for 10 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Newly diagnosed (previously untreated or currently receiving cancer treatment for the diagnosis that made the patient eligible for this study) with germ cell tumor, hepatoblastoma, medulloblastoma, neuroblastoma, osteosarcoma, or other malignancy
* Planning to receive a chemotherapy treatment regimen that includes a cumulative cisplatin dose ≥ 200 mg/m² with individual cisplatin doses to be infused over ≤ 6 hours
* Enrolled on hearing assessment clinical trial COG-ACCL05C1

  * Normal auditory results

PATIENT CHARACTERISTICS:

* Karnofsky performance status (PS) 50-100% (for patients > 16 years of age)
* Lansky PS 50-100% (for patients ≤ 16 years of age)
* Serum sodium normal
* Absolute granulocyte count > 1,000/mm³
* Platelet count > 100,000/mm³
* Creatinine clearance or radioisotope glomerular filtration rate ≥ 70mL/min OR serum creatinine between 0.4 and 1.7 mg/dL, based on age and gender
* Total bilirubin ≤ 1.5 times upper limit of normal (ULN) for age
* AST or ALT < 2.5 times ULN for age
* Not pregnant or nursing
* Negative pregnancy test (if patient has child-bearing capacity)
* Fertile patients must use effective contraception
* No known hypersensitivity to sodium thiosulfate or other thiol agents (e.g., amifostine trihydrate, N-acetylcysteine, MESNA, or captopril)

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior platinum-based chemotherapy (cisplatin or carboplatin)

  * Other prior chemotherapy allowed
* Prior cranial radiotherapy (e.g., for treatment of medulloblastoma) allowed provided normal hearing is documented after completion of radiotherapy and before enrollment and administration of cisplatin chemotherapy
* At least 6 months since prior hematopoietic stem cell transplantation.

  * No evidence of graft-versus-host disease
* No concurrent enrollment on another COG clinical trial for treatment of the cancer.

  * Concurrent enrollment on a non-COG clinical trial (e.g., Head start) allowed.
* Cranial irradiation after the completion of all systemic chemotherapy allowed provided post end-of-treatment audiometry is completed prior to beginning irradiation.
* Concurrent radiotherapy to extracranial sites allowed.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 131 (Actual)
Dates: Start 2008-06-23 (Actual); Primary Completion 2015-04-09 (Actual); Study Completion 2021-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David R. Freyer, DO, MS, Study Chair — Children's Hospital Los Angeles
Locations (76):
- United States (68):
  - UAB Comprehensive Cancer Center, Birmingham, Alabama
  - Arkansas Cancer Research Center at University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Childrens Hospital Los Angeles, Los Angeles, California
  - Southern California Permanente Medical Group, Los Angeles, California
  - Children's Hospital Central California, Madera, California
  - Rady Children's Hospital - San Diego, San Diego, California
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Yale Cancer Center, New Haven, Connecticut
  - Alfred I. duPont Hospital for Children, Wilmington, Delaware
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Lee Cancer Care of Lee Memorial Health System, Fort Myers, Florida
  - Nemours Children's Clinic, Jacksonville, Florida
  - University of Miami Sylvester Comprehensive Cancer Center - Miami, Miami, Florida
  - Florida Hospital Cancer Institute at Florida Hospital Orlando, Orlando, Florida
  - Nemours Children's Clinic - Orlando, Orlando, Florida
  - Nemours Children's Clinic - Pensacola, Pensacola, Florida
  - All Children's Hospital, St. Petersburg, Florida
  - St. Joseph's Cancer Institute at St. Joseph's Hospital, Tampa, Florida
  - Cancer Research Center of Hawaii, Honolulu, Hawaii
  - Mountain States Tumor Institute at St. Luke's Regional Medical Center, Boise, Idaho
  - University of Illinois Cancer Center, Chicago, Illinois
  - Saint Jude Midwest Affiliate, Peoria, Illinois
  - Riley's Children Cancer Center at Riley Hospital for Children, Indianapolis, Indiana
  - Blank Children's Hospital, Des Moines, Iowa
  - Holden Comprehensive Cancer Center at University of Iowa, Iowa City, Iowa
  - Kosair Children's Hospital, Louisville, Kentucky
  - Tulane Cancer Center Office of Clinical Research, Alexandria, Louisiana
  - Children's Hospital of New Orleans, New Orleans, Louisiana
  - National Naval Medical Center, Bethesda, Maryland
  - C.S. Mott Children's Hospital at University of Michigan Medical Center, Ann Arbor, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Helen DeVos Children's Hospital at Spectrum Health, Grand Rapids, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Children's Hospitals and Clinics of Minnesota - Minneapolis, Minneapolis, Minnesota
  - Masonic Cancer Center at University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - Children's Mercy Hospital, Kansas City, Missouri
  - Cardinal Glennon Children's Hospital, St Louis, Missouri
  - CCOP - Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Hackensack University Medical Center Cancer Center, Hackensack, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Herbert Irving Comprehensive Cancer Center at Columbia University Medical Center, New York, New York
  - SUNY Upstate Medical University Hospital, Syracuse, New York
  - Presbyterian Cancer Center at Presbyterian Hospital, Charlotte, North Carolina
  - Duke Cancer Institute, Durham, North Carolina
  - Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies and Children's Hospital, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Oklahoma University Cancer Institute, Oklahoma City, Oklahoma
  - Legacy Emanuel Children's Hospital, Portland, Oregon
  - Knight Cancer Institute at Oregon Health and Science University, Portland, Oregon
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Geisinger Cancer Institute at Geisinger Health, Danville, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Rhode Island Hospital Comprehensive Cancer Center, Providence, Rhode Island
  - Sanford Cancer Center at Sanford USD Medical Center, Sioux Falls, South Dakota
  - East Tennessee Children's Hospital, Knoxville, Tennessee
  - Driscoll Children's Hospital, Corpus Christi, Texas
  - Simmons Comprehensive Cancer Center at University of Texas Southwestern Medical Center - Dallas, Dallas, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Children's Hospital of The King's Daughters, Norfolk, Virginia
  - Virginia Commonwealth University Massey Cancer Center, Richmond, Virginia
  - Providence Cancer Center at Sacred Heart Medical Center, Spokane, Washington
  - St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Marshfield Clinic - Marshfield Center, Marshfield, Wisconsin
- Princess Margaret Hospital for Children, Perth, Western Australia, Australia
- Canada (7):
  - Children's and Women's Hospital of British Columbia, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - IWK Health Centre, Halifax, Nova Scotia
  - Hospital for Sick Children, Toronto, Ontario
  - Hopital Sainte Justine, Montreal, Quebec
  - Saskatoon Cancer Centre at the University of Saskatchewan, Saskatoon, Saskatchewan
  - Centre Hospitalier Universitaire de Quebec, Québec

REFERENCES:
- [Derived] Freyer DR, Chen L, Krailo MD, Knight K, Villaluna D, Bliss B, Pollock BH, Ramdas J, Lange B, Van Hoff D, VanSoelen ML, Wiernikowski J, Neuwelt EA, Sung L. Effects of sodium thiosulfate versus observation on development of cisplatin-induced hearing loss in children with cancer (ACCL0431): a multicentre, randomised, controlled, open-label, phase 3 trial. Lancet Oncol. 2017 Jan;18(1):63-74. doi: 10.1016/S1470-2045(16)30625-8. Epub 2016 Dec 1. PMID 27914822

RESULTS

PARTICIPANT FLOW:
Groups:
- STS Arm (Sodium Thiosulfate Treatment): Sodium thiosulfate treatment.
- Observation Arm: No sodium thiosulfate treatment.
Period: Overall Study
Arm/Group | STS Arm (Sodium Thiosulfate Treatment) | Observation Arm
Started | 65 | 66
Completed | 45 | 57
Not Completed | 20 | 9
Not completed — Adverse Event | 2 | 0
Not completed — Death | 1 | 0
Not completed — Physician Decision | 2 | 2
Not completed — Withdrawal by Subject | 5 | 1
Not completed — Premature discontinuation cisplatin | 5 | 4
Not completed — Radiation during protocol | 1 | 0
Not completed — Ineligibles | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | STS Arm (Sodium Thiosulfate Treatment) | Observation Arm | Total
Number analyzed (Participants) | 65 | 66 | 131
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 65 | 66 | 131
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 8.97 (5.93) | 8.39 (5.88) | 8.68 (5.89)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 24 | 51
  Male | 38 | 42 | 80
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 19 | 15 | 34
  Not Hispanic or Latino | 44 | 48 | 92
  Unknown or Not Reported | 2 | 3 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Black or African American | 7 | 10 | 17
  White | 44 | 41 | 85
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 11 | 12 | 23
Region of Enrollment [Number; unit: participants] — 1 patient of unknown origin in STS arm
  participants
    Canada | 8 | 4 | 12
    United States | 56 | 62 | 118

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Hearing Loss
Description: Hearing loss defined by comparing hearing sensitivity at follow up evaluation relative to baseline measurements using ASHA criteria.
Time Frame: 4 weeks after last dose of cisplatin
Population: 55 eligible patients enrolled on the observation Arm had complete audiometry data for evaluation; 49 eligible patients enrolled on the STS arm had complete data audiometry for evaluation.
Measure: Number; unit: Patients
Arm/Group | STS Arm (Sodium Thiosulfate Treatment) | Observation Arm
Number analyzed (Participants) | 49 | 55
Patients | 14 | 31

2. Secondary Outcome: Change in Hearing Thresholds For Key Frequencies at 500 hz
Description: Mean change in hearing threshold (post-pre) at 500 hz.
Time Frame: 4 weeks after last dose of cisplatin
Population: 38 eligible patients in the STS arm had paired audiometry at 500 hz; 45 patients in the observation arm had paired audiometry at 500 hz.
Measure: Mean (Standard Deviation); unit: Decibels
Arm/Group | STS Arm (Sodium Thiosulfate Treatment) | Observation Arm
Number analyzed (Participants) | 38 | 45
Decibels | -1.45 (5.80) | -1.11 (8.59)

3. Secondary Outcome: Change in Hearing Thresholds For Key Frequencies at 1000 hz
Description: Mean change in hearing threshold (post-pre) at 1000 hz.
Time Frame: 4 weeks after last dose of cisplatin
Population: 37 eligible patients in the STS arm had paired audiometry at 1000 hz; 47 patients in the observation arm had paired audiometry at 1000 hz.
Measure: Mean (Standard Deviation); unit: Decibels
Arm/Group | STS Arm (Sodium Thiosulfate Treatment) | Observation Arm
Number analyzed (Participants) | 37 | 47
Decibels | -0.676 (4.59) | -0.319 (8.99)

4. Secondary Outcome: Change in Hearing Thresholds For Key Frequencies at 2000 hz
Description: Mean change in hearing threshold (post-pre) at 2000 hz
Time Frame: 4 weeks after last dose of cisplatin
Population: 38 eligible patients in the STS arm had paired audiometry at 2000 hz; 47 patients in the observation arm had paired audiometry at 2000 hz.
Measure: Mean (Standard Deviation); unit: Decibels
Arm/Group | STS Arm (Sodium Thiosulfate Treatment) | Observation Arm
Number analyzed (Participants) | 38 | 47
Decibels | -1.18 (4.85) | 0.638 (12.7)

5. Secondary Outcome: Change in Hearing Thresholds For Key Frequencies at 4000 hz
Description: Mean change in hearing threshold (post-pre) at 4000 hz.
Time Frame: 4 weeks after last dose of cisplatin
Population: 38 eligible patients in the STS arm had paired audiometry at 4000 hz; 47 patients in the observation arm had paired audiometry at 4000 hz.
Measure: Mean (Standard Deviation); unit: Decibels
Arm/Group | STS Arm (Sodium Thiosulfate Treatment) | Observation Arm
Number analyzed (Participants) | 38 | 47
Decibels | 1.05 (7.09) | 9.58 (20.5)

6. Secondary Outcome: Change in Hearing Thresholds For Key Frequencies at 8000 hz
Description: Mean change in hearing threshold (post-pre) at 8000 hz.
Time Frame: 4 weeks after last dose of cisplatin
Population: 38 eligible patients in the STS arm had paired audiometry at 8000 hz; 42 patients in the observation arm had paired audiometry at 8000 hz.
Measure: Mean (Standard Deviation); unit: Decibels
Arm/Group | STS Arm (Sodium Thiosulfate Treatment) | Observation Arm
Number analyzed (Participants) | 38 | 42
Decibels | 9.73 (17.3) | 17.0 (24.7)

7. Secondary Outcome: Event-Free Survival (EFS)
Description: Proportion of patients event free at 4 years following enrollment. See EFS outcome measure description.
Time Frame: 4 years after enrollment
Population: 61 eligible patients were enrolled on the STS arm; 64 eligible patients were enrolled on the observation arm.
Measure: Number (95% Confidence Interval); unit: Percentage probability
Arm/Group | STS Arm (Sodium Thiosulfate Treatment) | Observation Arm
Number analyzed (Participants) | 61 | 64
Percentage probability | 53.7 [39.8 to 65.8] | 61.4 [48.0 to 72.3]

8. Secondary Outcome: Overall Survival (OS)
Description: Proportion of patients alive free at 4 years following enrollment. See OS outcome measure description.
Time Frame: 4 Years after enrollment
Population: 61 eligible patients were enrolled on the STS arm; 64 eligible patients were enrolled on the observation arm.
Measure: Number (95% Confidence Interval); unit: Percentage probability
Arm/Group | STS Arm (Sodium Thiosulfate Treatment) | Observation Arm
Number analyzed (Participants) | 61 | 64
Percentage probability | 69.6 [55.6 to 79.9] | 82.0 [68.4 to 90.1]

9. Secondary Outcome: Hearing Loss Among Patients Carrying/Not-carrying Two Key Gene Mutations (TPMT and COMT)
Time Frame: 4 weeks after the last dose of cisplatin
Population: Data was and never will be collected
Arm/Group | STS Arm (Sodium Thiosulfate Treatment) | Observation Arm (No Sodium Thiosulfate Treatment)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: Serious Adverse Events were reported on this study via the NCI AERS reporting system. Per protocol, no expedited reports were submitted for patients on Observation only arm of the study. Thus, no patients enrolled on the Observation arm of the trial were at risk for having a Serious Adverse Event reported.
Arm/Group | STS Arm (Sodium Thiosulfate Treatment) | Observation Arm
Serious Adverse Events (participants affected / at risk) | 21/59 | 0/0
Other Adverse Events (participants affected / at risk) | 51/59 | 57/64
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | STS Arm (Sodium Thiosulfate Treatment) (N=59) | Observation Arm (N=0)
Abdominal infection (Infections and infestations) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Acidosis (Metabolism and nutrition disorders) | 1 | 0
Alanine aminotransferase increased (Investigations) | 3 | 0
Anaphylaxis (Immune system disorders) | 1 | 0
Anemia (Blood and lymphatic system disorders) | 7 | 0
Anorexia (Metabolism and nutrition disorders) | 2 | 0
Anxiety (Psychiatric disorders) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 1 | 0
Conjunctivitis (Eye disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 0
Depressed level of consciousness (Nervous system disorders) | 1 | 0
Extrapyramidal disorder (Nervous system disorders) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 12 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 0
Hypoglycemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 1 | 0
Hypomagnesemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatremia (Metabolism and nutrition disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 0
Infections and infestations - Other, specify (Infections and infestations) | 3 | 0
Lymphocyte count decreased (Investigations) | 4 | 0
Mucositis oral (Gastrointestinal disorders) | 5 | 0
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 0
Neutrophil count decreased (Investigations) | 10 | 0
Oral pain (Gastrointestinal disorders) | 1 | 0
Pharyngeal stenosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Platelet count decreased (Investigations) | 8 | 0
Rectal pain (Gastrointestinal disorders) | 1 | 0
Reversible posterior leukoencephalopathy syndrome (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 2 | 0
Typhlitis (Gastrointestinal disorders) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Weight loss (Investigations) | 1 | 0
White blood cell decreased (Investigations) | 8 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | STS Arm (Sodium Thiosulfate Treatment) (N=59) | Observation Arm (N=64)
Abdominal infection (Infections and infestations) | 0 | 1
Acidosis (Metabolism and nutrition disorders) | 1 | 1
Alanine aminotransferase increased (Investigations) | 7 | 9
Allergic reaction (Immune system disorders) | 5 | 3
Anemia (Blood and lymphatic system disorders) | 23 | 36
Anorexia (Metabolism and nutrition disorders) | 2 | 4
Anxiety (Psychiatric disorders) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 4 | 5
Blood bilirubin increased (Investigations) | 1 | 0
Bone infection (Infections and infestations) | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Catheter related infection (Infections and infestations) | 0 | 3
Chills (General disorders) | 2 | 0
Colitis (Gastrointestinal disorders) | 0 | 1
Confusion (Psychiatric disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 3
Device related infection (Infections and infestations) | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Enterocolitis infectious (Infections and infestations) | 0 | 1
Esophageal infection (Infections and infestations) | 0 | 1
Esophageal pain (Gastrointestinal disorders) | 0 | 1
Esophageal ulcer (Gastrointestinal disorders) | 1 | 0
Esophagitis (Gastrointestinal disorders) | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 19
GGT increased (Investigations) | 3 | 1
Hearing impaired (Ear and labyrinth disorders) | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 1
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 0
Hypermagnesemia (Metabolism and nutrition disorders) | 1 | 3
Hypernatremia (Metabolism and nutrition disorders) | 7 | 4
Hypertension (Vascular disorders) | 1 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 4 | 2
Hypokalemia (Metabolism and nutrition disorders) | 15 | 13
Hypomagnesemia (Metabolism and nutrition disorders) | 2 | 2
Hyponatremia (Metabolism and nutrition disorders) | 7 | 4
Hypophosphatemia (Metabolism and nutrition disorders) | 12 | 7
Hypotension (Vascular disorders) | 1 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Infections and infestations - Other, specify (Infections and infestations) | 3 | 9
Infusion related reaction (General disorders) | 0 | 2
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1 | 0
Leukoencephalopathy (Nervous system disorders) | 1 | 0
Lymphocyte count decreased (Investigations) | 2 | 9
Middle ear inflammation (Ear and labyrinth disorders) | 0 | 1
Mucositis oral (Gastrointestinal disorders) | 3 | 4
Nausea (Gastrointestinal disorders) | 3 | 3
Neutrophil count decreased (Investigations) | 39 | 51
Otitis media (Infections and infestations) | 1 | 0
Pain (General disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Paronychia (Infections and infestations) | 0 | 1
Penile infection (Infections and infestations) | 0 | 1
Perineal pain (Reproductive system and breast disorders) | 1 | 0
Peripheral motor neuropathy (Nervous system disorders) | 1 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0
Pharyngitis (Infections and infestations) | 1 | 0
Platelet count decreased (Investigations) | 30 | 39
Sepsis (Infections and infestations) | 0 | 2
Sinusitis (Infections and infestations) | 1 | 1
Skin infection (Infections and infestations) | 1 | 2
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 | 0
Upper respiratory infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 1
Vomiting (Gastrointestinal disorders) | 3 | 3
Weight loss (Investigations) | 1 | 0
White blood cell decreased (Investigations) | 30 | 42
Wound infection (Infections and infestations) | 0 | 1

LIMITATIONS AND CAVEATS:
Data was and never will be collected for Outcome Measure #9, Hearing Loss Among Patients Carrying/Not-carrying Two Key Gene Mutations (TPMT and COMT).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Must obtain prior Sponsor approval.